CLINICAL TRIAL: NCT06973590
Title: Effects of Low-intensity Resistance Training With Blood Flow Restriction and Transcutaneous Electrical Nerve Stimulation on Lower Limb Motor Function in People With Stroke
Brief Title: Blood Flow Restriction and Transcutaneous Electrical Nerve Stimulation on Motor Function in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Prof., The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025_BFR+TENS_STROKE
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Chronic Stroke
Keywords: blood flow restriction; transcutaneous electrical nerve stimulation; stroke; low-intensity resistance training
MeSH Terms: conditions — Stroke | interventions — Blood Flow Restriction Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LIRT + BFR + TENS (Experimental): All subjects will receive 60-minute sessions of LIRT with both actual BFR and actual TENS intervention, 3 sessions per week for 6 weeks.
  Interventions: Device: Blood flow restriction (BFR); Device: Transcutaneous electrical nerve stimulation (TENS); Behavioral: Low-intensity resistance training (LIRT)
- LIRT + sham BFR + TENS (Sham Comparator): All subjects will receive 60-minute sessions of LIRT with simulated BFR and actual TENS, 3 sessions per week for 6 weeks.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS); Device: Sham blood flow restriction (Sham-BFR); Behavioral: Low-intensity resistance training (LIRT)
- LIRT + BFR + sham TENS (Sham Comparator): All subjects will receive 60-minute sessions of LIRT with actual BFR and simulated TENS, 3 sessions per week for 6 weeks.
  Interventions: Device: Blood flow restriction (BFR); Device: Sham transcutaneous electrical nerve stimulation (Sham-TENS); Behavioral: Low-intensity resistance training (LIRT)
- LIRT + sham BFR + sham TENS (Placebo Comparator): All subjects will receive 60-minute sessions of LIRT with simulated BFR and simulated TENS, 3 sessions per week for 6 weeks.
  Interventions: Device: Sham blood flow restriction (Sham-BFR); Device: Sham transcutaneous electrical nerve stimulation (Sham-TENS); Behavioral: Low-intensity resistance training (LIRT)

INTERVENTIONS:
Device: Blood flow restriction (BFR) — BFR implementation involves an automated restriction band (SmartCuffs 4.0) positioned at the proximal region of the affected lower extremity, calibrated to 50% of the individual's lower limb occlusion pressure (LOP). The pressure system remains inflated throughout active training phases and is systematically deflated during inter-exercise intervals.
  Arms: LIRT + BFR + TENS; LIRT + BFR + sham TENS
Device: Transcutaneous electrical nerve stimulation (TENS) — TENS will be delivered to the anterior thigh region of the paretic leg using a 120z Dual-Channel TENS Unit (ITO Physiotherapy & Rehabilittaion, Co, Ltd, Tokyo, Japan). The TENS stimulation will be at 100 Hz, with 0.2 ms square pulses at an intensity of twice the sensory threshold (defined as the minimum intensity at which subject reported feeling a tingling sensation and below the motor threshold as indicated by the absence of muscle twitching.
  Arms: LIRT + BFR + TENS; LIRT + sham BFR + TENS
Device: Sham blood flow restriction (Sham-BFR) — Sham BFR implementation involves an automated restriction band (SmartCuffs 4.0) positioned at the proximal region of the affected lower extremity, calibrated to 50% of the individual's lower limb occlusion pressure (LOP). But the pressure system remains deflated throughout active training and resting phases.
  Arms: LIRT + sham BFR + TENS; LIRT + sham BFR + sham TENS
Device: Sham transcutaneous electrical nerve stimulation (Sham-TENS) — Sham TENS will be delivered to the anterior thigh region of the paretic leg using a 120z Dual-Channel TENS Unit (ITO Physiotherapy & Rehabilittaion, Co, Ltd, Tokyo, Japan). The TENS stimulation will be at 100 Hz, with 0.2 ms square pulses at an intensity of twice the sensory threshold (defined as the minimum intensity at which subject reported feeling a tingling sensation and below the motor threshold as indicated by the absence of muscle twitching. But the stimulator will only be applied for the first and last 30 seconds.
  Arms: LIRT + BFR + sham TENS; LIRT + sham BFR + sham TENS
Behavioral: Low-intensity resistance training (LIRT) — The LIRT protocol utilizes 20% of one-repetition maximum (1-RM) as the standardized training load. LIRT including leg extensions, leg presses, and load-bearing squats focused on the affected limb. Each resistance exercise consists of 3 sets of 20 repetitions with rest intervals.

SUMMARY:
Stroke commonly results in persistent leg impairments that limit mobility and reduce quality of life. This study investigates whether combining low-intensity resistance training with blood flow restriction (LIRT-BFR) and transcutaneous electrical nerve stimulation (TENS) can effectively improve leg function in stroke survivors.

Participants with chronic stroke will be randomly assigned to one of four intervention groups: 1) LIRT with simulated BFR and simulated TENS; 2) LIRT with actual BFR and simulated TENS; 3) LIRT with simulated BFR and actual TENS; 4) LIRT with both actual BFR and actual TENS. The resistance training utilizes 20% of each participant's maximum lifting capacity. For blood flow restriction, an automated pressure cuff (SmartCuffs 4.0) will be placed on the upper portion of the affected leg, inflated to 50% of the individual's occlusion pressure during exercises and deflated during rest periods. TENS therapy delivers controlled electrical impulses through electrodes positioned on the anterior thigh.

Each 60-minute session includes a 10-minute warm-up followed by 40 minutes of targeted resistance exercises (leg extensions, leg presses, and weight-bearing squats) and concludes with 10 minutes of stationary cycling. The resistance protocol involves 3 sets of 20 repetitions with standardized rest intervals between sets and exercises. Participants will attend three sessions weekly for six weeks.

Assessments will be conducted at baseline, midpoint (3 weeks), completion (6 weeks), and follow-up (1 month post-intervention). The primary outcome measure is the Fugl-Meyer Assessment for Lower Extremity function, with secondary measures including muscle strength, stiffness, balance, mobility, walking capacity, and gait parameters. To understand the underlying mechanisms, we will measure muscle oxygenation using near-infrared spectroscopy, evaluate muscle structure via ultrasound, and monitor physiological responses including heart rate variability and perceived exertion for safety monitoring.

DETAILED DESCRIPTION:
Stroke often leads to persistent lower-limb impairments, limiting functional recovery and quality of life. Low-intensity resistance training with blood flow restriction (LIRT-BFR) has shown promise in improving muscle function in healthy populations, but its effects in stroke rehabilitation remain underexplored. Additionally, while BFR and electrical stimulation have been beneficial for pain relief and muscle activation, the impact of combining BFR with transcutaneous electrical nerve stimulation (TENS) in stroke patients remains unknown. The objectives of this study is to evaluate whether a multi-mode exercise rehabilitation training program of LIRT-BFR and TENS can restore lower extremity strength, mobility, and quality of life.

In this randomized controlled trial, chronic stroke patients will be allocated to one of four groups: 1) LIRT + sham BFR + sham TENS, 2) LIRT + BFR + sham TENS, 3) LIRT + sham BFR + TENS, and 4) LIRT + BFR + TENS. The LIRT protocol utilizes 20% of one-repetition maximum (1-RM) as the standardized training load. BFR implementation involves an automated restriction band (SmartCuffs 4.0) positioned at the proximal region of the affected lower extremity, calibrated to 50% of the individual's lower limb occlusion pressure (LOP). The pressure system remains inflated throughout active training phases and is systematically deflated during inter-exercise intervals. TENS application targets the anterior thigh region.

The intervention protocol comprises a structured 60-minute session beginning with a 10-minute preparatory warm-up, followed by 40 minutes of targeted resistance exercises including leg extensions, leg presses, and load-bearing squats focused on the affected limb, concluding with 10 minutes of aerobic cycling. Each resistance exercise consists of 3 sets of 20 repetitions with rest intervals. The assessments will be conducted at baseline, mid-intervention (3 weeks), post-intervention (6 weeks), and follow-up (1 month post-completion).

The primary outcome measure will be the Fugl-Meyer Assessment Lower Extremity (FMA-LE) score, and secondary outcome measures including muscle strength, stiffness, balance, functional mobility, walking capacity, gait speed, etc. To elucidate the underlying mechanisms, the study will use near-infrared spectroscopy (NIRS) to assess muscle oxygenation and hemodynamics, ultrasound for muscle morphology, and exercise measures like heart rate variability (HRV) and rating of perceived exertion (RPE) for safety consideration.

ELIGIBILITY:
Inclusion Criteria:

1. are between 50 and 80 years of age;
2. have had a single stroke more than 6 months and less than 15 years;
3. have at least 5 degrees of active ankle dorsiflexion in the antigravity position;
4. are able to walk 10 m independently, with or without a walking aid;
5. are able to score 6 or higher out of 10 on the abbreviated mental test;
6. have no skin allergies (e.g. redness or itchiness after application of the electrical stimulation pads) to electrical stimulation or electrodes;
7. are able to follow instructions and give informed consent.

Exclusion Criteria:

1. presence of other comorbidities like varicose veins, peripheral neuropathy, cancer, musculoskeletal injury, lower limb peripheral edema, post-surgical swelling, open wounds, or on a medication that increases blood clotting risk;
2. resting blood pressure ≥ 160/100 mmHg even after taking medications, cardiovascular comorbidity, heart failure, unstable angina, by-pass surgery, a pacemaker;
3. administration of botulinum toxin in the lower limb at least 6 months prior to training;
4. history of epilepsy, cochlear implants, any type of deep brain stimulator and metal implants in the head or neck;
5. currently not participating in resistance training or high-intensity or long duration cardiovascular exercise;
6. lack the ability to feel pain (because of paralysis), or other subjects who cannot complain of discomfort.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Lower Extremity (FMA-LE) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  FMA-LE is used to evaluate the lower extremity motor control, including reflexes, voluntary control of isolated movement and coordination. The scale score ranging from 0 to 34, with 17 items and ordinal scoring from 0 to 2. A higher score indicates a better lower extremity motor control.

SECONDARY OUTCOMES:
Paretic ankle dorsiflexor/plantarflexor strength | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The paretic ankle dorsiflexor/plantarflexor strength (in kilograms) is measured with a Nicholas hand-held dynamometer (model 01165, Lafayette Instrument Company, Lafayette, IN) in supine lying position. The muscle strength will be measured twice. The average strength of the 2 trials will be recorded. A higher value indicated a better paretic ankle dorsiflexor/plantarflexor strength.
Knee extension strength | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  Knee extension strength is measured using a Cybex isokinetic dynamometer in isometric mode. Participants will be seated with their back supported and hips flexed at 90°. The axis of rotation of the dynamometer will be aligned with the lateral femoral epicondyle, and the resistance pad will be secured just proximal to the malleoli on the anterior aspect of the leg. The test will be conducted with the knee positioned at 90° of flexion. Following familiarization with the procedure, participants will perform three maximal voluntary isometric contractions, each held for 5 seconds with a 60-second rest period between attempts. The average peak torque value from the three trials will be recorded in Newton-meters (Nm). Higher values indicate greater knee extension strength.
10-Meter Walk Test (10MWT) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The subject will be asked to walk 10 meter in a comfortable speed. The completion time will be records by stopwatch. The test will be repeated for 2 times. The completion time will be averaged. The shorter the completion time, the better performance is.
Timed 'Up and Go' test (TUG) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The TUG is used to measure the functional mobility. Each subject will be required to rise from a chair with armrests, walk 3 m forward, turn around, return to the chair and sit down. The time taken to complete this task will be measured in seconds with a stopwatch. Each condition will be repeated for 2 times. The completion time will be averaged.
Gait Parameters (via GAITRite) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  Gait parameters will be assessed using the GAITRite system (CIR system, Inc., Havertown, Pennsylvania), a pressure-sensitive mat that automatically captures spatiotemporal gait characteristics. Participants will walk at their self-selected comfortable pace along the instrumented walkway.
Berg Balance Scale (BBS) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  BBS is a 14-item objective measure that assesses static balance and fall risk in adult patients. Items include tasks such as sitting to standing, standing unsupported, transfers, reaching, turning 360 degrees, and single-leg stance. Each item is scored from 0-4 points (0=unable to perform, 4=independent), with a maximum total score of 56 points. Higher scores indicate better balance.
Limits of Stability (LOS) Test | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The Limits of Stability (LOS) test quantifies participants' ability to intentionally shift their center of gravity (COG) to their stability limits without losing balance using Bertec Balance Advantage System (Bertec Corporation, Columbus, OH, USA). Participants stand on a force plate and shift their weight to move a cursor on a screen toward 8 targets arranged in a circular pattern at their theoretical limits of stability (100% LOS). Key parameters measured reaction time (RT) , movement velocity (MVL), directional control (DCL), endpoint excursion (EPE), maximum excursion (MXE). Higher scores indicate better dynamic balance control, except for reaction time where lower scores are better.
Weight bearing distribution | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  Weight bearing distribution will be assessed using the Bertec Balance Advantage System (Bertec Corporation, Columbus, OH, USA). Participants will stand barefoot on the dual force plate platform with feet positioned at shoulder width and arms resting at their sides. The system's integrated software will measure vertical ground reaction forces under each foot to calculate the percentage of weight distribution between the affected and unaffected lower extremities. Weight bearing measurements will be conducted under four conditions: (1) relaxed standing balance, (2) squat position at 30° knee flexion, (3) squat position at 60° knee flexion, (4) squat position at 90° knee flexion. For each squat position, participants will be instructed to maintain the position for 10 seconds while a handrail will be available for safety but not for weight support.
Ultrasound muscle thickness | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  Muscle thickness will be evaluated using B-mode ultrasonography with a 5-12 MHz linear-array transducer. Measurements will be performed with participants in a supine position after 10 minutes of rest to allow fluid redistribution. Standard anatomical landmarks will be used to ensure measurement consistency: Rectus Femoris at 50% of the distance between the anterior superior iliac spine and the superior border of the patella; Vastus Lateralis at 2/3 of the distance from the anterior superior iliac spine to the lateral side of the patella; Tibialis Anterior at 30% of the distance from the lateral condyle of the tibia to the lateral malleolus; and Gastrocnemius Medialis at 30% of the distance from the popliteal crease to the lateral malleolus. The transducer will be positioned perpendicular to the muscle surface with minimal pressure to avoid tissue compression. Three consecutive images will be captured for each muscle, and muscle thickness will be measured as the perpendicular distance

CONTACTS AND LOCATIONS:
Overall Officials: Shamay NG, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No